Development and Implementation of an Infusion Monitoring System to Prevent Phlebitis, Infiltration, and Extravasation in the Intensive Care Unit

08.08.2025

## INFORMED CONSENT FORM

This form was prepared by the faculty members of the Department of Fundamentals of Nursing, Faculty of Health Sciences, Karadeniz Technical University. The title of the research is "Development and Implementation of an Infusion Monitoring System to Prevent Phlebitis, Infiltration, and Extravasation in the Intensive Care Unit." This study aims to develop an infusion monitoring system for the early detection of complications associated with peripheral intravenous catheters and to evaluate its effectiveness. Data will be collected using the "Clinical Monitoring Form," "Patient Information Form," and "Complication Monitoring Form." All information provided during our interviews will be used solely for this research, and personal information will be kept strictly confidential. Furthermore, participants' names will not be included in the research report when presenting the study results. The duration of the study is 19 months. During this period, you are expected to answer the questions regarding your health status as accurately as possible to ensure the reliability of the research findings. Below are the contact details of the researcher you can reach within the scope of the study.

Participant's Statement: I, ......., have read all the explanations in the Informed Consent Form. I received both written and verbal information about the research mentioned above, including its purpose and subject, from the researcher named below. I voluntarily agree to participate in the study, and I understand that I can withdraw from the study at any time, with or without stating a reason. I accept to participate in this research of my own free will, without any pressure or coercion.

| free will, without any pressure or coercion. |
|--------------------------------------------------------------|
| Participant's Full Name (Legal representative if necessary): |
| Signature: Address (Phone number if applicable): |
| Date (day/month/year):/ |
| Researcher Providing the Explanation – Full Name: |
| Address: Phone number: Date (day/month/year):/ |
| Signature: |